CLINICAL TRIAL: NCT05880355
Title: Multimodality Cardiovascular Imaging for the Translation of Therapies for Vascular Activation After MI
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Lindner, MD, Professor of Medicine, Vice Chief for Research, Cardiovascular Division, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR230183
Record Dates: First submitted 2023-05-04; First posted 2023-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — dapansutrile

STUDY DESIGN:
Intervention Model Description: Randomized, single blind study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapansutrile (Experimental): Subjects randomized to receive oral dapnsutrile
  Interventions: Drug: Dapansutrile
- Control (Placebo Comparator): Subjects randomized to receive oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapansutrile — Oral inhibitor of NLRP3
  Arms: Dapansutrile
Other: Placebo — Non-active placebo
  Arms: Control

SUMMARY:
Subjects with urgently reperfused type I myocardial infarction (MI) will be recruited and randomized to receive either placebo or the oral inflammasome (NLRP3) inhibitor dapansutrile. The primarily outcome measure will be carotid plaque volume change over 6 months; secondary outcome measures will be plaque inflammatory activity and coronary microvascular function.

ELIGIBILITY:
Inclusion Criteria:

* Acute type I myocardial infarction (NSTEMI or STEMI)
* Reperfusion therapy planned or performed within prior 48 hrs
* Carotid or femoral artery plaque at baseline, or carotid intima media thickness >1.5 mm

Exclusion Criteria:

* Type II MI
* Failed primary PCI or need for emergent bypass surgery
* Severe heart failure (NYHA class IV)
* Life-threatening complication of MI (myocardial rupture, ischemic VSD, papillary muscle rupture)
* Refractory ventricular arrhythmias
* Allergy to dapansutril, OLT177, or drugs in the same class
* Co-morbidity limiting 6 month survival
* Active malignancy or recent malignancy with any systemic anti-cancer treatment
* Active infection
* Use of immunosuppressive medications or immunodeficiency disorder
* Neutropenia (ANC <2,000)
* Moderate or severe renal impairment (GFR <30 ml/min)
* Recent stroke (within previous 3 months)
* Allergy to ultrasound enhancing agents or polyethylene glycol
* Pregnancy or breastfeeding

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Remote plaque volume | 6 months
  Carotid artery plaque volume change by ultrasound measured by 3D ultrasound. Outcome units will be cm3 averaged for bilateral carotid arteries.

SECONDARY OUTCOMES:
Plaque inflammation | 3 months
  Carotid artery plaque inflammatory activity by PET-CT. Units will be SVU averaged bilaterally for a region-of-interest over the carotid bifurcation.
Coronary microvascular function | 3 months
  Coronary microvascular reactivity by myocardial contrast echo (MCE) quantitative perfusion imaging. The primary endpoint unit will be coronary microvascular flux rate reserve (regadenoson stress: rest ratio).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided